CLINICAL TRIAL: NCT06387134
Title: Study on the Therapeutic Effect of Lifei Xiaoji Wan on Lung Adenocarcinoma in the Early Stage of Ground Glass Nodule (Ia Stage) and Its Effect on Tumor Microenvironment
Brief Title: Lifei Xiaoji Wan Treatment's of Early-stage NSCLC and Its Impact on the Tumor Microenvironment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCM for early-stage LUAD
Record Dates: First submitted 2024-04-17; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Early Stage Lung Adenocarcinoma
Keywords: early stage lung adenocarcinoma; tumor microenvironment; ground glass nodule

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): The patients in the trial group received routine Western medicine treatments, and oral Lifei Xiaoji Wan (10 pills/time,3 times/day).
  Interventions: Drug: Lifei Xiaoji Wan
- control group (Placebo Comparator): The patients in the control group received routine Western medicine treatments.
  Interventions: Drug: Conventional treatment with Western medicine

INTERVENTIONS:
Drug: Lifei Xiaoji Wan — The Lifei Xiaoji Wan consists of ginseng, blackhead,rhubarb, aster, forehu, and thin on.
  Arms: trial group
Drug: Conventional treatment with Western medicine — Recommended treatment protocols for patients with Stage Ia NSCLC in the "Chinese Society of Oncology Branch of Lung Cancer Clinical Diagnosis and Treatment Guidelines for Lung Cancer (2021 edition)" and the "Chinese Society of Clinical Oncology (CSCO) Non-small Cell Lung Cancer Diagnosis and Treatment Guidelines 2021".
  Arms: control group

SUMMARY:
This study evaluated the relationship between the clinical efficacy, histopathological changes and tumor microenvironment of the pharmacopharmacologic Lifei Xiaoji Wan in the treatment of early stage lung adenocarcinoma, and improved high-level clinical evidence and action targets for the prevention and treatment of early stage lung cancer by traditional Chinese medicine

DETAILED DESCRIPTION:
Lung cancer is a malignant tumor with the highest morbidity and mortality. The microenvironment of tumor plays an important role in its occurrence and development.Traditional Chinese medicine has great advantages in the prevention and treatment of ground glass pulmonary nodules, but there is a lack of high-level clinical evaluation evidence and precise mechanism of action.Lifei Xiaoji Wan is a prescription based on the theory of "gas accumulation causing cancer". It has good curative effect in treating non-small cell lung cancer.

In this study, a single-center randomized controlled study was used to set up a treatment group and a control group to observe and evaluate the clinical efficacy of Lifeixiaoji pills on patients with early stage lung adenocarcinoma of ground glass nodules. Flow cytometry, PCR array and multiple fluorescence immunofluorescence were used to detect the tumor microenvironment in lung cancer tissues. To investigate the effect of Lifeixiaoji pill on tumor microenvironment and its mechanism of action on early lung adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* It met the diagnostic criteria of non-small cell lung cancer and was confirmed by pathology, cytology and other relevant examinations.
* Preoperative thin-slice CT showed pure ground glass pulmonary nodules with a size of 10mm-30mm. Intraoperative and postoperative pathology indicated adenocarcinoma, and the tumor stage (TNM) was stage Ia.
* Age: 18-75 years old
* Expected survival >5 years
* Informed consent and sign informed consent

Exclusion Criteria:

* Patients who have undergone surgery
* Patients with serious dysfunction of heart, liver, lung, kidney and other important organs
* Patients with mental illness who were unable to complete the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Quality of Life Scale (FACT-L) | There are 36 items in the scale, and each item is scored as 0~4 points, with a total score range of 0-144 points (minimum: 0 points; maximum value: 144 points).Higher dimensions and total scores indicate higher.Change from baseline at month 1 and 2.
  FACT-L scale was used to record the patients' physiological status, social/family status, emotional status and functional status
TCM symptoms and syndromes | Change from baseline at month 1 and 2.
  The evaluation was carried out according to the standard of TCM syndrome of lung cancer in Guiding Principles for Clinical Research of New Chinese Medicine
Evaluation of tumor efficacy using RECIST criteria to measure changes in tumor body | Every 1 month, assessed up to 2 months, CT was collected for imaging analysis and measurement.RECIST criteria for tumor efficacy evaluation:The extent of growth or shrinkage of the target lesion (unit: mm).
  The changes of tumor body and lesion were observed and the therapeutic effect on tumor was evaluated

SECONDARY OUTCOMES:
Tumor markers：CEA | Every 1 month, assessed up to 2 months.
  Tumor marker CEA levels.
Tumor markers：CA211 | Every 1 month, assessed up to 2 months.
  Tumor marker CA211 levels.
Tumor markers：squamous cell carcinoma antigen | Every 1 month, assessed up to 2 months.
  Tumor marker squamous cell carcinoma antigen levels.
Complete blood count: white blood cells | Every 1 month, assessed up to 2 months.
  white blood cells levels.
Complete blood count: haemoglobin | Every 1 month, assessed up to 2 months.
  haemoglobin levels.
Complete blood count: Platelet | Every 1 month, assessed up to 2 months.
  Platelet levels.
Liver function tests: ALT | Every 1 month, assessed up to 2 months.
  Liver function tests ALT levels.
Liver function tests: AST | Every 1 month, assessed up to 2 months.
  Liver function tests AST levels.
Renal function tests: BUN | Every 1 month, assessed up to 2 months.
  Renal function tests BUN levels.
Renal function tests: Cr | Every 1 month, assessed up to 2 months.
  Renal function tests Cr levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Mingli Zhao, Zhengzhou, China

IPD SHARING:
Plan to Share IPD: No